CLINICAL TRIAL: NCT06481046
Title: Treatment of Rotator Cuff Tears With Platelet Rich Plasma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Use of PRP does not require a registered clinical trial
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015RC
Record Dates: First submitted 2020-10-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tendinitis
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Dual injections of PRP - 4 ml injected into each location. The first injection was into the supraspinatus tendon insertion critical zone and bursal area with the patient seated. The second injection was performed with the patient prone into the glenohumeral intra-articular space under the supraspinatus tendon at, or just proximal to, the superior equator of the humeral head.
  Interventions: Biological: Platelet Rich Plasma (PRP)

INTERVENTIONS:
Biological: Platelet Rich Plasma (PRP) — Platelet Rich Plasma (PRP) prepared from patient blood, spun twice to concentrate platelets. 45 cc of initial blood resulting in 4cc of injectable PRP.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of dual platelet rich plasma (PRP) injections into the rotator cuff insertion and the area of the tendon proximal to the insertion.

DETAILED DESCRIPTION:
Patients who have rotator cuff pathology as established by clinical exam and confirmed with MRI and have failed activity modification, will be enrolled in this study. They will receive dual platelet rich plasma (PRP) injections, one into the rotator cuff insertion and one into the area of the tendon proximal to the insertion, in one treatment session. PRP will be prepared through a double spin technique to create two 4 cc doses for injection. Patients will evaluated at 6 months, 1 year and two years for improvement in symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff pathology established by exam
* Rotator cuff pathology confirmed with MRI.
* Failure to improve with activity modification and physical therapy
* Willingness to stop all NSAID medication

Exclusion Criteria:

* Additional significant shoulder pathology seen on xray or MRI including: severe arthritis, significant superior labrum anterior postierior (SLAP) Type II lesions and intra-articular loose bodies.
* Shoulder surgery within 6 months.
* Presence of full thickness rotator cuff tears in patients amenable to surgical repair.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2015-01-25 (Actual); Study Completion 2015-01-25 (Actual)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand Score (Quick-DASH) | change from baseline to 6 months
  Quick-DASH questionnaire consists of 11 questions which are each scored 1-5. The scoring ranges from 0 for best to 100 for worst outcomes.
Quick Disabilities of the Arm, Shoulder and Hand Score (Quick-DASH) | change from baseline to 12 months
  Quick-DASH questionnaire consists of 11 questions which are each scored 1-5. The scoring ranges from 0 for best to 100 for worst outcomes.
Quick Disabilities of the Arm, Shoulder and Hand Score (Quick-DASH) | change from baseline to 24 months
  Quick-DASH questionnaire consists of 11 questions which are each scored 1-5. The scoring ranges from 0 for best to 100 for worst outcomes.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for pain | change from baseline to 6 months
  The Visual Analog Scale is a single question about current pain level. Scoring ranges from 0 which is no pain to 100 which is worst possible pain.
Visual Analog Scale (VAS) for pain | change from baseline to 12 months
  The Visual Analog Scale is a single question about current pain level. Scoring ranges from 0 which is no pain to 100 which is worst possible pain.
Visual Analog Scale (VAS) for pain | change from baseline to 24 months
  The Visual Analog Scale is a single question about current pain level. Scoring ranges from 0 which is no pain to 100 which is worst possible pain.
Global Improvement | change from baseline to 6 months
  Global improvement is a single question about percent improved compared to before treatment where 0 is not improved and 100 is completely improved.
Global Improvement | change from baseline to 12 months
  Global improvement is a single question about percent improved compared to before treatment where 0 is not improved and 100 is completely improved.
Global Improvement | change from baseline to 24 months
  Global improvement is a single question about percent improved compared to before treatment where 0 is not improved and 100 is completely improved.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — Illinois Sportsmedicine and Orthopaedic Centers
Locations (1):
- Illinois Sportsmedicine and Orthopaedic Centers, Glenview, Illinois, United States

IPD SHARING:
Plan to Share IPD: No